CLINICAL TRIAL: NCT03126890
Title: Investigation of the Correlation Between Plasma Concentration of Linezolid Antibiotic and Treatment Response and Adverse Reactions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201610008RINB
Record Dates: First submitted 2016-11-30; First posted 2017-04-25 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Myelosuppression; Lactic Acidosis; Peripheral Neuropathy
Keywords: Pharmacokinetics,adverse events; Linezolid; Therapeutic drug monitoring; Myelosuppression; Lactic acidosis; Peripheral neuropathy
MeSH Terms: conditions — Acidosis, Lactic; Peripheral Nervous System Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood for drug concentration monitoring
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Linezolid TDM (prospective): Adult patients received linezolid at NTUH. This prospective cohort study will draw blood from every patient to measure the linezolid blood concentration. After blood concentration analysis by high pressure liquid chromatography (HPLC), the investigator will report the concentration to clinicians and dose adjustment is judged by clinician (not the investigators).
- Linezolid observation (retrospective): Adult patients received linezolid at NTUH.

SUMMARY:
Linezolid is the second line agent in the treatment of MRSA and PRSP infections, and it is also the drug of choice for VRE infections. It can be an alternative option against multidrug resistant tuberculosis and non-tuberculosis mycobacterium. However, Patients who receive more than 2 weeks of treatment duration and who have renal dysfunction or severe cirrhosis may prone to experience anemia, thrombocytopenia, and leukopenia. Long-term use may also result in lactic acidosis, peripheral neuropathy and optic neuropathy due to mitochondrial toxicity. Thus, this study will analysis the medical charts in National Taiwan University Hospital (NTUH) from 2011 to 2016 to get the population demographics who use linezolid and analysis the occurrence rate of myelosuppression, neuropathy and lactic acidosis. Simultaneously, the investigators also use therapeutic drug monitoring (TDM) to prospectively evaluate the association of linezolid blood concentration and clinical efficacy and safety. The result of this study will provide physicians more information to prevent concentration-dependent adverse effects.

DETAILED DESCRIPTION:
The increasing resistance of methicillin-resistant Staphylococcus aureus (MRSA), vancomycin-resistant enterococci (VRE), and penicillin-resistant Streptococcus pneumoniae (PRSP) has caused significant medical issue. With limited antimicrobial agents available, it has been an increasing challenge in infection control and disease treatment. Linezolid is the second line antibiotics in the treatment of MRSA and PRSP infections, and it is also the drug of choice for VRE infections. It can be an alternative against multidrug resistant tuberculosis and non-tuberculosis mycobacterium. Linezolid has almost 100% of bioavailability. It has excellent tissue penetration. It metabolized via non-enzymatic oxidation. Two major metabolites, aminoethoxyacetic acid (chemical name) and hydroxyethyl glycine (chemical name), are final forms before excreted through kidneys. Even though the manufacturer does not recommend dosing adjustment for patients with renal or hepatic dysfunction, recent studies demonstrated accumulation of linezolid and 2 metabolites in the body. Patients who receive more than 2 weeks of treatment duration and who have renal dysfunction or severe cirrhosis may present higher plasma linezolid concentration. Patients may experience anemia, thrombocytopenia, and leukopenia under long-term use of linezolid. However, there is lack of study on lactic acidosis, peripheral neuropathy, and optic neuropathy due to mitochondrial toxicity.

This study has two parts. This study will analysis the medical charts in NTUH from 2011 to 2016 to get the population demographics who use linezolid and the occurrence rate of myelosuppression, neuropathy and lactic acidosis. Then, followed by a prospective study which aim is to monitor the plasma peak and trough concentration of linezolid (total and free drug) and 2 metabolites by different sample collecting method (plasma, dry blood spot; DBS). If clinical necessity, the investigators may also monitor tissue fluid concentration. Clinical response and toxicity were monitored by liquid chromatography (LC) analysis. The investigators plan to evaluate the association between plasma concentration and toxicity including bone marrow suppression, peripheral neuropathy, and lactic acidosis. It is important to determine if dose adjustment in patients with renal and/or hepatic dysfunction is required. Simultaneously, the investigators want to develop DBS method which can ease patients' uncomfortable sense and simplify the drug monitor process. The result of this study will provide physicians more information to prevent concentration-dependent adverse effects.

ELIGIBILITY:
Retrospective study 1. Adults (age > 20 year old) with linezolid treatment (oral or intravenous) in National Taiwan University hospital medical charts record from 2011 to 2016. 2. Patients with linezolid treatment for 3 days or above Prospective study

1. Adults (age > 20 year old) are going to start with linezolid treatment (oral or intravenous) due to gram positive infection, multidrug resistant - tuberculosis (MDR-TB) or nontuberculous mycobacterium (NTM) infection.
2. Keeping follow up in National Taiwan University Hospital

Exclusion Criteria:

Retrospective study 1. Patients without baseline complete blood count (CBC) data (RBC or Hb, WBC, platelet) before linezolid treatment. Prospective study

1. Patients with severe disease status (assess by clinicians) might die within 2 days or treatment duration less than 2 days

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with oral or intravenous linezolid
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-11-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical efficacy | Observation periods: entire linezolid treatment course until 30 days after the completion of treatment, loss of follow up, death or December 2020 (up to 4 years).
  Clinical efficacy definition:
  Cure: biological eradication or clinical improvement. (Biological eradication: Eradication of bacterial culture prior to study drug) (Clinical improvement: White blood cell (WBC), C reactive protein (CRP) back to normal range (WBC: 3500 - 9000/mm3; CRP: < 1 mg/dL) or without sepsis symptom (body temperature, pulse, heart rate returned to normal))
  Intermittent cure: same bacteria culture positive (with same minimum inhibitory concentration (MIC) data) within 2 weeks after linezolid treatment ends.
  Failure: persistent bacteria culture after linezolid treatment or unresolved clinical sign and symptoms.
  Indeterminate outcome: loss of follow up or discontinue linezolid due to adverse drug reaction
Safety - thrombocytopenia | Observation periods: entire linezolid treatment course until resolution of side effect, loss of follow up, death or December 2020 (up to 4 years).
  Definition of thrombocytopenia: platelet count < 100,000/mm3 and platelet count of < 75% of the baseline counts.
Safety - anemia | Observation periods: entire linezolid treatment course until resolution of side effect, loss of follow up, death or December 2020 (up to 4 years).
  Definition of anemia: Hemoglobin (Hb) < 10 g/dL and Hb level of < 75% of the baseline level.
Safety - leukopenia | Observation periods: entire linezolid treatment course until resolution of side effect, loss of follow up, death or December 2020 (up to 4 years).
  Definition of leukopenia: WBC count < 3000/mm3 and WBC count of < 50% of baseline count.
Safety - lactic acidosis | Observation periods: entire linezolid treatment course until resolution of side effect, loss of follow up, death or December 2020 (up to 4 years).
  Definition of lactic acidosis:
  1. Definite lactic acidosis: lactic acid > 4 mmol/L and blood potential of hydrogen (pH) value < 7.35
  2. Probable lactic acidosis: lactic acid > 4 mmol/L without or not achieved pH value data
Safety - peripheral neuropathy | Observation periods: entire linezolid treatment course until resolution of side effect, loss of follow up, death or December 2020 (up to 4 years).
  Definition of peripheral neuropathy (PN):
  1. Definite PN: with nerve conduction velocity test (+)
  2. Probable PN: patient reported symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Wen Lin, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Test2, Taiwan